CLINICAL TRIAL: NCT04374916
Title: Evaluation of a New Predictive Test of Preterm Birth in Case of Threatened Preterm Labor
Acronym: PREMAQUICK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7353
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Threatened Preterm Labor; Preterm Delivery
Keywords: Threatened preterm labor; Preterm Delivery; Preterm birth; IGFBP-1
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partosure® test + Premaquick® test (Experimental): All patients will have the same 2 tests.
  Interventions: Device: Premaquick®; Device: PARTOSURE®

INTERVENTIONS:
Device: Premaquick® — Vaginal secretions are collected prior to any vaginal or endovaginal ultrasound examination to avoid false positives, with the nylon swab provided with the test (placed in the posterior fornix of the vagina for 10 seconds).Then the samples are tested with the Premaquick test. Results are obtained in 10 minutes.
Device: PARTOSURE® — An immunochromatographic test wich determines the qualitative in vitro detection of placental alpha microglobulin-1 (PAMG-1) in cervico-vaginal secretions.

SUMMARY:
Threatened preterm labor (TPL) is defined by cervical changes and regular and painful uterine contractions occurring between 24 and 36 + 6 weeks of gestation that may or may not lead to premature labor and delivery. There is no reliable way to predict preterm delivery.

The study's hypothesis is that the Premaquick® test can improve the prediction of preterm delivery.

The investigators also want to compare this test with the Partosure® (Placental alpha microglobulin-1) test.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 years (with no upper age limit)
* Patient affiliated to a social security health regime
* Between 24 and 33 + 6 weeks of gestation (amenorrhea)
* Singleton pregnancy
* Patient with a TPL: Uterine contractions during the last 24 hours felt by the patient, painful or not, and cervix less than or equal to 25 mm on endovaginal ultrasound
* Having signed an informed consent form

Exclusion Criteria:

* Twin pregnancy
* Sexual intercourse less than 24 hours from inclusion
* Cervical cerclage
* Abundant metrorrhagia
* Premature rupture of membranes
* Pre-eclampsia
* Congenital malformation
* Presence of a placenta previa
* Pelvic examination in the previous 24 hours (compared to inclusion)
* Patient under guardianship, curatorship or safeguard of justice
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care under duress

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-08-25 (Estimated); Study Completion 2022-08-25 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the occurrence of a premature delivery within 7 days after patient's inclusion. | The outcome measure is assessed at visit 2 (day 7), 7 days after the inclusion visit.

SECONDARY OUTCOMES:
Collection of the occurrence of a premature delivery within 7 days of inclusion, then calculation of specificity, positive and negative predictive values. | At visit 2, Day 7 (7 days after inclusion visit V0)
Collection of the occurrence of a premature delivery on Day 2 and Day 14 following the inclusion, then calculation of the sensitivities, specificities, positive and negative predictive values. | At visit 1, Day 2 (2 days after inclusion visit ) and D14 (14 days after inclusion visit )
Collection of the number of invalid results requiring restarting the Premaquick test. | At the Inclusion visit Visit 0 (Day 0)
Collection of premature deliveries at different times (2, 7 and 14 days after inclusion visit), then comparison of the sensitivities and specificities of the two tests at different times. | At visit 1 (Day 2) - Visit 2 (Day 7) and after end of research visit (Day 14)
a new calculation algorithm to predict the risk of preterm delivery, based on the results observed in this study. | At visit 1 (Day 2) - Visit 2 (Day 7) and after end of research visit (Day 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided